CLINICAL TRIAL: NCT00164918
Title: Role of Routine Nasogastric Decompression After Subtotal Gastrectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2004.311
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Cancer of Stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Enteral Nutrition

INTERVENTIONS:
Device: nasogastric tube

SUMMARY:
The aim of the study is to evaluate whether subtotal gastrectomy without post-operative nasogastric decompression is better in terms of early post-operative bowel function and chest complication.

DETAILED DESCRIPTION:
Nasogastric decompression is an intra-operative routine in most of the time to facilitate exposure of operative field during elective subtotal gastrectomy, but whether it should be retained post-operatively is controversial. Nasogastric decompression helps to drain the gastric remnant in case there is edema around the gastrojejunostomy, ileus and delayed gastric emptying, which can theoretically relieve nausea and abdominal distension. Besides, it may help decrease diaphragmatic splintage and hence decrease chance of chest infection if ileus occurs. However, nasogastric intubation could cause patient discomfort; also it has been shown that it would cause gastroesophageal reflux which may be associated with chest complication. There have been studies showing that routine post-operative nasogastric decompression is not necessary for gastrectomy in general, but the role in subtotal gastrectomy for stomach cancer is not well defined.

ELIGIBILITY:
Inclusion Criteria:All patients suffering from carcinoma of stomach, decided for operation

* subtotal, D1/D2 dissection
* palliative resection

Exclusion Criteria:

* actively bleeding tumor
* perforation of tumor
* patient present with gastric outlet obstruction
* combine organ excision
* known diabetes with nephropathy

Min Age: 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2004-09

PRIMARY OUTCOMES:
Bowel function and related symptoms early post-op

CONTACTS AND LOCATIONS:
Overall Officials: Enders K.W. Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Surgical Ward, Prince of Wales Hospital, Hong Kong, China